CLINICAL TRIAL: NCT04468217
Title: Evaluation of an Alternative Method of Obtaining Viral RNA for the Detection of SARS-CoV-2 Virus Using PCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neurognos (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-02
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: COVID; SARS-CoV2; Corona Virus Infection
Keywords: SARS-CoV-2; Diagnostics; RNA Extraction; COVID
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with positive test to SARS-COV2: Employees of critical services companies and healthcare workers with a positive test to SARS-COV2.
  Interventions: Diagnostic Test: Obtainment of nasopharyngeal, oropharyngeal, buccal, nasal and saliva samples
- Subjects with negative test to SARS-COV2: Employees of critical services companies and healthcare workers with a negative test to SARS-COV2.
  Interventions: Diagnostic Test: Obtainment of nasopharyngeal, oropharyngeal, buccal, nasal and saliva samples

INTERVENTIONS:
Diagnostic Test: Obtainment of nasopharyngeal, oropharyngeal, buccal, nasal and saliva samples — Each patient will undergo a sample collection where two nasopharyngeal samples will be obtained, one of them with lysis buffer as the transport medium and the other with the AAA-Safe solution as the transport medium. Oropharyngeal, buccal, nasal, and salivary samples will also be obtained using AAA-Safe as the transport medium

SUMMARY:
The current coronavirus disease pandemic has posed a problem and a challenge for health systems globally. In the framework of a pandemic, a diagnosis is a key tool in containing and monitoring disease outbreaks.

In this pandemic, the qPCR technique has become vitally important in virus detection, due to its wide detection and quantification range, and the high levels of sensitivity and specificity it presents. The methodology for diagnosing coronavirus by qPCR requires the prior extraction of viral genetic material, which is carried out using commercial kits created for this purpose. Currently, the high demand for supplies to carry out this technique has generated reagent shortage problems, including commercial kits for the extraction of viral genetic material.

This research aims to evaluate a solution called AAA-Safe and its method, developed to optimize the diagnostic process, eliminating and replacing the viral RNA extraction stage. We hope that this alternative can be implemented in any molecular diagnostic laboratory, in order to speed up the delivery of a fast and safe diagnosis.

DETAILED DESCRIPTION:
This analytical and non-interventional study will evaluate the performance of a new workflow for the detection of SARS-CoV-2 viral RNA from samples of nasopharyngeal, oropharyngeal, buccal, nasal and saliva mucosa using as transport medium the propietary AAA-Safe solution, in 150 volunteers in two different locations. The first sampling location will be held in a private clinic, where healthcare professionals will be enrolled. The second sampling location will be held at an essential services company, where samples will be taken by employees who voluntarily want to participate in the study.

All volunteers will be informed of all aspects of this protocol and must sign an informed consent before there participation. All the information associated with the samples requested will be duly anonymized in order to protect the identity of the volunteers.

The extracted samples will be processed and analyzed to obtain the detection limit of the diagnostic flow by implementing the developed solution and to establish the clinical performance in terms of sensitivity and specificity of the technique.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Volunteer able to understand and sign the informed consent
* Healthcare professionals
* Essential services company workers

Exclusion Criteria:

* Older than 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups can be identified within the study population:
  * The first group are health professionals (nurses, doctors, kinesiologists, etc.) who are working in healthcare centers during the current pandemic.
  * The second group are employees of an essential services company.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of an alternative method of obtaining viral RNA for the detection of SARS-CoV-2 virus in nasopharyngeal samples. | 3 months
  Two workflows for the detection of SARS-CoV-2 will be compared:
  Gold Standard: Obtaining nasopharyngeal sample in validated transport medium, RNA extraction by columns and qPCR.
  Alternative method: Obtaining nasopharyngeal sample in AAA-Safe proprietary transport medium, alternative method of extraction and qPCR.

SECONDARY OUTCOMES:
Evaluation of an alternative method of obtaining viral RNA for the detection of SARS-CoV-2 virus in oropharyngeal, nasal, buccal and saliva samples | 3 months
Establish a sample bank of nasopharyngeal, oropharyngeal, nasal, buccal and saliva mucosa for future analytical validations of new solutions associated with the detection of the SARS-CoV-2 virus. | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorio Neurognos, Santiago, Providencia, Chile

IPD SHARING:
Plan to Share IPD: Undecided